CLINICAL TRIAL: NCT05509608
Title: Evaluation of an Electroretinogram Sensor
Brief Title: Evaluating a New Sensor That Measures the Health of the Retina in Normally-sighted Subjects
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: RetMap, Inc (Industry)
Collaborators: University of Illinois at Chicago (Other); Illinois College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RMEFDA2022
Record Dates: First submitted 2022-07-14; First posted 2022-08-22 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-09

CONDITIONS: Electrode Site Reaction
Keywords: Electroretinogram; Sensor; Retina; Contact lens; Electrode; Efficacy; Feasibility

STUDY DESIGN:
Intervention Model Description: This study is structured with two Arms (Aims).
  For the first Arm (Aim 1) of this study, subjects (n=10) wear two ERG sensors, a new contact lens electrode and an FDA approved contact lens electrode, one after the other. The signal quality of the recorded ERG responses obtained with each sensor will be compared. Comparison of signal quality will help in assessing the functionality of the new contact lens electrode.
  For the second Arm (Aim 2) of this study, subjects (n=10) will wear the two ERG sensors at the same time, one in each eye. After 20, 40 and 60 minutes of wear, each eye will be examined for irritation using standard clinical scales. Observing for ocular irritation will help determine the effect of the devices on the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Electroretinogram Signal Quality (Experimental): Electroretinogram Signal Quality: This Arm will participate in a comparative study using two ERG sensors, one commercially available electrode and one seeking FDA approval (RM Electrode). This will be done by performing standard ERG test protocols with both electrodes worn one at a time, in one eye (random order) in ten healthy (normally-sighted) adult subjects.
  Interventions: Device: RM Electrode; Device: ERG Jet Electrode
- Ocular Irritation (Experimental): Ocular Irritation: Ten healthy (normally-sighted) adult subjects will wear the RM Electrode in one eye and a commercially available electrode in the other eye for a total of 60 minutes, in 20-minute sessions with short breaks in between. The eyes will be evaluated for irritation (standard clinical grading scales for bulbar redness, limbal redness, tarsal redness, and slit-lamp examination of corneal staining) after each 20-minute interval.
  Interventions: Device: RM Electrode; Device: ERG Jet Electrode

INTERVENTIONS:
Device: RM Electrode — The RM Electrode is a corneal ERG electrode. The distinguishing features of the RM electrode are that it is a soft contact lens with a recessed electrode (i.e. no metal electrode makes direct contact with the eye). The RM Electrode also has an integral speculum to hold the wearer's eye lids open. The electrode is designed for superior positional stability on the eye during testing. These features work together to improve ERG signal quality.
Device: ERG Jet Electrode — The ERG Jet electrode is an FDA approved, commercially available corneal ERG electrode.

SUMMARY:
The primary purpose of this study is to evaluate the ability of a new contact lens electrode to record a measurable electroretinogram (ERG). ERG sensors in various forms have been in common clinical use for more than 50 years. The ERG sensor that is the subject of this study is the RM Electrode, developed by RetMap, Inc. (project sponsor). The RM Electrode is not yet approved by the FDA. The RM Electrode will be compared to other commercially available electrode

The first Aim of the present study is to compare the functionality of the RM Electrode and other commercially available electrodes. Following standard ERG test protocols, responses will be recorded from ten healthy (normally-sighted) adult subjects using both electrodes (used in random order). The signal quality of the ERG responses obtained from both contact lens electrodes will be compared. Signal quality will be determined by measuring ERG signal amplitudes and calculating signal-to-noise ratios (SNR). Signal-to-noise ratios will be used to establish substantial equivalence. ERG test results will not be used to determine the effect of the devices on the participants.

The second Aim of the present study is to evaluate the risk of ocular irritation caused by use of the RM Electrode compared to other commercially available electrodes. A typical ERG test session lasts 20 minutes. Ten healthy (normally-sighted) adult subjects will wear the RM Electrode on one eye and a commercially available electrode on the other eye, for a total of 60 minutes, in 20-minute sessions with short breaks in between. To determine the effect of the devices on the participants, the eyes will be evaluated for irritation.

ELIGIBILITY:
Inclusion Criteria:

* Persons 18 and over.

Exclusion Criteria:

* Pregnant woman
* Individuals with existing diagnosis for any retinal disease, ocular surgery (including refractive surgery such as Lasik) within the past six months, corneal ulcers, or any noticeable ocular irritation on the study day.
* Non-English speaking persons may not enroll.
* Persons who may respond negatively to flashing lights in the eye will be excluded, or excused from the study if enrolled and the negative response is revealed during the study.

Excluded or Vulnerable Populations:

* No vulnerable populations are expected to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Arm1: ERG signal quality, including peak amplitudes, noise levels, and signal to noise ratios. | Up to 24 weeks
  Signals recorded from both contact lens electrode will be evaluated for a-wave and b-wave peak amplitudes, signal power, noise power and signal-to-noise ratios.
Arm 2: Ocular irritation using clinical grading scales | Up to 24 weeks
  Slit-lamp examination and standard clinical grading scales for bulbar redness, limbal redness, tarsal redness, and corneal staining (fluorescein).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hyde, MD/PhD, Principal Investigator — UIC Department of Ophthalmology & Visual Sciences; Michael Chaglasian, OD, Principal Investigator — Illinois College of Optometry
Locations (2):
- United States (2):
  - UIC Department of Ophthalmology & Visual Sciences, Chicago, Illinois
  - Illinois College of Optometry, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCulloch DL, Marmor MF, Brigell MG, Hamilton R, Holder GE, Tzekov R, Bach M. ISCEV Standard for full-field clinical electroretinography (2015 update). Doc Ophthalmol. 2015 Feb;130(1):1-12. doi: 10.1007/s10633-014-9473-7. Epub 2014 Dec 14. PMID 25502644
- [Background] Hoffmann MB, Bach M, Kondo M, Li S, Walker S, Holopigian K, Viswanathan S, Robson AG. ISCEV standard for clinical multifocal electroretinography (mfERG) (2021 update). Doc Ophthalmol. 2021 Feb;142(1):5-16. doi: 10.1007/s10633-020-09812-w. Epub 2021 Jan 25. PMID 33492495